CLINICAL TRIAL: NCT02086838
Title: Comparison Between Iron Supplementation Using Total Dose Infusion and Oral Routes for Treatment of Iron Deficiency Anemia in Pregnancy
Brief Title: Iron Supplementation Using Total Dose Infusion and Oral Routes for Treatment of Iron Deficiency Anemia in Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Lecturer of Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9020058
Record Dates: First submitted 2014-03-12; First posted 2014-03-13 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Treatment of Iron Deficiency Anemia in Pregnancy
Keywords: Iron deficiency anemia; Pregnancy; Iron therapy
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theragran Hematinic, oral iron, 120 mg elemental iron/ (Active Comparator): pregnant women taking 60 mg elemental iron twice per day (120 mg/day) using iron tablets (Theragran Hematinic)® SmithKline Beecham, Egypt an affiliated co. to GlaxoSmithKline. Adherence to the treatment will be monitored by asking the women to bring back the empty packs and mark the consumption of tablets on calendar.
  Interventions: Drug: Theragran Hematinic
- low molecular weight iron dextran, total dose infusion (Active Comparator): Pregnant women taking elemental iron in the form of low molecular weight dextran complex intravenously as a total dose infusion (T.D.I) using iron dextran ampules (Cosmofer)R pharmacosmos Denmark (Inspire Pharma Egypt). Patients selected for parental iron will be admitted as day cases in the hospital in a single visit. The required dose has to be individually adapted according to the total iron deficit which is dependent on the patient's body weight and hemoglobin status. Total iron dose (mg) = weight (kg) X Hemoglobin deficit {target Hemoglobin (g/l)- Actual Hemoglobin (g/l)} X 0.24 + 500 mg.
  Interventions: Drug: low molecular weight iron dextran

INTERVENTIONS:
Drug: Theragran Hematinic
  Arms: Theragran Hematinic, oral iron, 120 mg elemental iron/
Drug: low molecular weight iron dextran
  Other Names: Cosmofer
  Arms: low molecular weight iron dextran, total dose infusion

SUMMARY:
Evaluate the effect of iron supplementation using oral routes in comparison with total dose infusion of low molecular weight iron dextran in iron deficiency anemia during pregnancy.

DETAILED DESCRIPTION:
Patients will be allocated to two groups of 106 each and to insure that everyone has the chance of participation, randomization will be guided by table of random numbers All women recruited in the study will be given 100 mg mebendazole tablets twice daily for 3 days for de-worming and 500 micro gram folic acid daily till the end of the study The required dose will be individually adapted according to the total iron deficit which is dependent on the patient's body weight and hemoglobin status Total iron dose (mg) = weight (kg) X hemoglobin deficit {target hemoglobin (g/l)- Actual hemoglobin (g/l)} X 0.24 + 500 mg The total iron dose needed will be calculated by formula rounded to nearest multiple of 100 Group I includes pregnant women taking 60 mg elemental iron twice per day (120 mg/day) using iron tablets (Theragran Hematinic)® Smith-Kline Beecham, Egypt an affiliated co. to Glaxo Smith-Kline, according to the WHO guidelines for IDA control Group II includes pregnant women taking elemental iron in the form of low molecular weight dextran complex intravenously as a total dose infusion (T.D.I) using iron dextran ampules (Cosmofer)R Pharmacosmos Denmark (Inspire Pharma Egypt) Inclusion criteria

* Maternal age 20-35 years old.
* Singleton pregnancy between 16 - 24 weeks
* Iron deficiency anemia with average hemoglobin ranging from 7-9 g/dL at the onset of the study

Exclusion criteris

* Extremes of reproductive age (less than 20 years old or more than 35 years old).
* Patients with multiple pregnancies.
* Anemia not linked to iron deficiency.
* Allergy to iron derivatives.
* Any medical disorder like diabetes or tuberculosis (TB), viral hepatitis cirrhosis, cardiovascular disease, renal disease, autoimmune disease, suspected acute infection, cancer.
* Those who had received parenteral iron treatment earlier within 3 months before the start of the study.
* Any obstetric complicating factors like pregnancy induced hypertension (PIH).
* Patients with history of chronic blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 20-35 years old.
* Singleton pregnancy between 16 - 24 weeks.
* Iron deficiency anemia with average hemoglobin ranging from 7-9 g % at the onset of the study.

Exclusion Criteria:

* Extremes of reproductive age (less than 20 years old or more than 35 years old).
* Patients with multiple pregnancies.
* Anemia not linked to iron deficiency.
* Allergy to iron derivatives.
* Any medical disorder like diabetes or tuberculosis (TB), viral hepatitis cirrhosis, cardiovascular disease, renal disease, autoimmune disease, suspected acute infection, cancer.
* Those who had received parenteral iron treatment earlier within 3 months before the start of the study.
* Any obstetric complicating factors like pregnancy induced hypertension.
* Patients with history of chronic blood loss.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who have been successfully treated | up to 8 weeks from comleting treatment
  The proportion of patients who have been successfully treated as evidenced by a hemoglobin concentration of > 10.5 g% after 8 weeks from completing treatment (oral or total iron dose infusion therapy).

SECONDARY OUTCOMES:
Number of participants with adverse effects | up to 8 weeks after completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S. Sweed, MD, Principal Investigator — AinShams University; Hazem M. Sammour, Professor, Study Director — AinShams University; Abdel-Latif G. El-Kholy, Ass. Prof., Principal Investigator — AinShams University; Eman M. El-Garhi, M.B.B.Ch., Principal Investigator — El Galaa Teaching Hospital
Locations (1):
- Maternity Hospital, Faculty of Madicine, AinShams University, Cairo, Egypt